CLINICAL TRIAL: NCT04790981
Title: Motor Imagery Training is an Effective Rehabilitation Program in Treatment of Children With Cerebellar Mutism
Brief Title: Effect of Motor Imagery Training on Ataxic Children After Medulloblastoma Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Saeed Alsakhawi, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/ 012/001935
Record Dates: First submitted 2021-02-26; First posted 2021-03-10 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Cerebellar Ataxia
MeSH Terms: conditions — Cerebellar Ataxia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- selected physical therapy program group (Active Comparator): The Control group received the selected physical therapy program for one hour, three times weekly for three successive months including facilitation of balance and protective reactions from standing position, standing on one leg, weight shifting from standing, squat to standing, strengthening exercises for trunk muscles and for upper and lower extremities musculatures, gait training activities for correction of gait pattern
  Interventions: Other: physical thertapy training
- motor imaginary training and selected physical therapy program group (Active Comparator): The study group received the selected physical therapy program for one hour, three times weekly for three successive months in addition to motor imagery program for 30 minutes as the following.
  Each child shown a video of 5 minutes of illustrating normal movements while the child resting in semi-reclined sitting in quiet room in front the screen. Children then asked to close their eyes and imagine practicing the task like the illustrative video. Repetition of the exercises depend on the children ranging from 5 to 10 repetitions per exercise
  Interventions: Other: motor imaginary training

INTERVENTIONS:
Other: motor imaginary training — Each child shown a video of 5 minutes of illustrating normal movements while the child resting in semi-reclined sitting in quiet room in front the screen. Children then asked to close their eyes and imagine practicing the task like the illustrative video. Repetition of the exercises depend on the children ranging from 5 to 10 repetitions per exercise.
  Arms: motor imaginary training and selected physical therapy program group
Other: physical thertapy training — The Control group received the selected physical therapy program for one hour, three times weekly for three successive months including facilitation of balance and protective reactions from standing position, standing on one leg, weight shifting from standing, squat to standing, strengthening exercises for trunk muscles and for upper and lower extremities musculatures, gait training activities for correction of gait pattern including.
  Arms: selected physical therapy program group

SUMMARY:
Background: after resection of medulloblastoma in children they suffer from signs and symptoms of ataxia which impedes their activities of daily living.

purpose: to investigate the effect motor imagery training on balance, severity of ataxia and gait parameters on children after resection of medulloblastoma.

Methods: Fifty children surfing from cerebellar ataxia after medulloblastoma resection were selected from tumors hospital of Cairo University, their age ranged from seven to nine years old, they were randomly assigned into two matched control and study groups. The control groups received the selected physical therapy program while, the study group received motor imaginary training in addition to the selected physical therapy program. Both groups were evaluated by ataxic rating scale, pediatric berg balance scale and kinematic gait analysis by kinovea software.

DETAILED DESCRIPTION:
Motor imagery is an effective method to enhance motor performance applied in rehabilitation programs it did not impose a physical load on patients, was confirmed through clinical evidence from meta-analysis. Motor imagery means thinking in motor task with executing it to activate motor cortical areas as 25% of the brain neurons are mirror neurons and fire by thinking.

ELIGIBILITY:
Inclusion Criteria:

* The children had signs of ataxia
* loss of balance
* able to understand and execute test instructions
* the children are in the follow up period after medulloblastoma resection.

Exclusion Criteria:

* medically unstable
* visual impairment
* increased intracranial pressure
* any other neuromuscular diseases.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Severity of ataxia | 3 months
  Scale for the Assessment and Rating of Ataxia to determine the degree of ataxia. It has eight items that yield a total score of 0 (no ataxia) to 40 (most severe ataxia)
Pediatric berg balance scale | 3 months
  to assess balance all children were assessed by the 14 items of the scale including sitting to standing, standing to sitting, transfers, standing unsupported, sitting unsupported, stand with eye closed, stand with feet together, standing with one foot in front, standing on one foot, turning 360 degrees, turning to look behind, retrieving object from floor, placing alternate foot on stool, and reaching forward without stretched arm. The total scale score range from 0 to 56.
step length (cm) | 3 months
  Kinematic gait analysis: Temporo-spatial gait variables were measured using a 2D motion analysis system. The kin markers were placed at greater trochanter, lateral femoral epicondyle, lateral malleolus and 5th metatarsal head. The tripod fixed with a video camera placed at 3 meters away from the walkway and focused on the middle part to record around 3 gait cycles of sagittal plane motion. The Kinovea software version 8.15.0 used to measure step length, stride length, cadence and walking speed. The measurement involved one trial of walking at the preferred gait speed along the 4 meters walkway
step width (cm) | 3 months
  Kinematic gait analysis: Temporo-spatial gait variables were measured using a 2D motion analysis system. The kin markers were placed at greater trochanter, lateral femoral epicondyle, lateral malleolus and 5th metatarsal head. The tripod fixed with a video camera placed at 3 meters away from the walkway and focused on the middle part to record around 3 gait cycles of sagittal plane motion. The Kinovea software version 8.15.0 used to measure step length, stride length, cadence and walking speed. The measurement involved one trial of walking at the preferred gait speed along the 4 meters walkway
foot angle (degree) | 3 months
  Kinematic gait analysis: Temporo-spatial gait variables were measured using a 2D motion analysis system. The kin markers were placed at greater trochanter, lateral femoral epicondyle, lateral malleolus and 5th metatarsal head. The tripod fixed with a video camera placed at 3 meters away from the walkway and focused on the middle part to record around 3 gait cycles of sagittal plane motion. The Kinovea software version 8.15.0 used to measure step length, stride length, cadence and walking speed. The measurement involved one trial of walking at the preferred gait speed along the 4 meters walkway
Cadence (steps/min) | 3 months
  Kinematic gait analysis: Temporo-spatial gait variables were measured using a 2D motion analysis system. The kin markers were placed at greater trochanter, lateral femoral epicondyle, lateral malleolus and 5th metatarsal head. The tripod fixed with a video camera placed at 3 meters away from the walkway and focused on the middle part to record around 3 gait cycles of sagittal plane motion. The Kinovea software version 8.15.0 used to measure step length, stride length, cadence and walking speed. The measurement involved one trial of walking at the preferred gait speed along the 4 meters walkway
Gait velocity (cm/sec) | 3 months
  Kinematic gait analysis: Temporo-spatial gait variables were measured using a 2D motion analysis system. The kin markers were placed at greater trochanter, lateral femoral epicondyle, lateral malleolus and 5th metatarsal head. The tripod fixed with a video camera placed at 3 meters away from the walkway and focused on the middle part to record around 3 gait cycles of sagittal plane motion. The Kinovea software version 8.15.0 used to measure step length, stride length, cadence and walking speed. The measurement involved one trial of walking at the preferred gait speed along the 4 meters walkway

CONTACTS AND LOCATIONS:
Overall Officials: Reham Alsakhawi, Ph.D., Principal Investigator — Assistant Professor, Faculty of Physical Therapy, Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data from participants will be made available
Supporting Information: Study Protocol
Time Frame: 12 months after study completion
Access Criteria: data access requests will be reviewed by an external independent review panel. requestor will be required to sign a data access agreement